CLINICAL TRIAL: NCT05542979
Title: A Randomized, Double-blind, Placebo-controlled Phase Ib Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Multiple-dose HH-003 Injection in Treatment Naïve Participants With HBeAg-positive Chronic HBV Infection
Brief Title: A Study to Evaluate the Safety, Tolerability of HH-003 Injection in Participants With Chronic Hepatitis B Virus Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Huahui Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HH0031802
Record Dates: First submitted 2022-09-11; First posted 2022-09-16 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Chronic HBV Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HH-003 Group (Experimental)
  Interventions: Drug: HH-003 injection
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HH-003 injection — HH-003 injection is administrated via I.V. infusion
  Arms: HH-003 Group
Drug: Placebo — Placebo is administrated via I.V. infusion
  Arms: Placebo Group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, multiple-ascending dose phase Ib study of HH-003 injection, which is a monoclonal antibody targeting Hepatitis B virus. This study aims to evaluate the safety, tolerability and pharmacokinetics of HH-003 injection in treatment-naive participants chronically infected with hepatitis B virus.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 45 years old
* Body weight ≥ 45 kg for men and ≥ 40 kg for women, and 18 kg/m^2≤BMI≤28 kg/m^2
* Positive serum HBsAg or HBV DNA for at least 6 months,or previous liver biopsy results confirm the Hepatitis B
* HBeAg positive, and 2000 IU/mL<HBsAg<100,000 IU/mL
* Have not received interferon treatment before, and have not received nucleotide/nucleoside analogue treatment within 6 months prior to Screening

Exclusion Criteria:

* Positive test for hepatitis C antibody (HCV-Ab), treponema pallidum antibody (TP-Ab), or anti-HIV antibody (HIV-Ab)
* Hemoglobin <100 g/L, platelets <100,000/mm^3 (100×10^9/L), absolute neutrophils count <1,500/mm^3 (1.5×10^9/L)
* Serum albumin <35 g/L, international normalized ratio (INR)>1.5; serum creatinine >115 μmol/L, Glomerular Filtration Rate (GFR) <70 mL/min/1.73m^2(calculated by Modification of Diet in Renal Disease (MDRD) formula); uric acid>540 μmol/L; triglyceride>3.5mmol/L
* Participants with a history of alcoholic liver disease, moderate or higher nonalcoholic fatty liver disease, autoimmune liver disease, Gilbert syndrome or other hereditary liver disease, drug-induced liver disease and other chronic liver diseases
* Participants with a history of progressive liver fibrosis (eg: liver cirrhosis diagnosed by liver histopathological examination, or esophagogastric varices diagnosed by endoscopy)
* Participants with confirmed or suspected decompensated HBV cirrhosis with complications of ascites, hepatic encephalopathy, gastroesophageal variceal bleeding, and Child-Pugh score of B~C, or with primary liver cancer
* Alpha Fetoprotein (AFP) >50 ng/ml at screening or the suspected malignant liver mass indicated by imaging
* Any previous or current malignant neoplasms
* Breast-feeding or pregnant females
* Participants who are not suitable to participate in this trial per the Investigator's judgment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From the first dose of study drug until Day 57
Peak concentration (Cmax) | From predose to Day 113
Area under the drug-time curve (AUC0-2W） | From predose to Day 113
Area under the drug-time curve (AUClast) | From predose to Day 113
Area under the drug-time curve (AUCinf) | From predose to Day 113

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Beijing Ditan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Friendship Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Youan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Mengchao Hepatobiliary Hospital Of Fujian Medical University, Fuzhou, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou, Henan
  - Henan Infectious Disease Hospital(The Sixth Peoples Hospital Of Zhengzhou), Zhengzhou, Henan
  - The First Hospital of Jilin University, Changchun, Jilin
  - Yanbian University Hospital(Yanbian Hospital), Yanji, Jilin
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - The First Affiliated Hospital,Zhejiang University School Of Medicine, Hangzhou, Zhejiang